CLINICAL TRIAL: NCT02362672
Title: A Phase 3 Double-Blind, Placebo-Controlled Study to Assess the Efficacy, Safety, and Tolerability of NKTR-181 in Opioid-Naive Subjects With Moderate to Severe Chronic Low Back Pain
Brief Title: Efficacy and Safety Study of NKTR-181 in Opioid-Naive Subjects With Low Back Pain
Acronym: SUMMIT-07
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Nektar Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 14-181-07
Record Dates: First submitted 2015-02-09; First posted 2015-02-13 (Estimated); Results first posted 2020-09-16 (Actual); Last update posted 2020-09-16 (Actual); Status verified 2020-09

CONDITIONS: Low Back Pain; Chronic Pain
MeSH Terms: conditions — Low Back Pain; Chronic Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- NKTR-181 (Experimental): NKTR-181 twice daily (BID) tablets
  Interventions: Drug: NKTR-181 BID tablets
- Placebo (Placebo Comparator): Placebo to match NKTR-181 twice daily (BID) tablets
  Interventions: Drug: Placebo to match NKTR-181 BID tablets

INTERVENTIONS:
Drug: NKTR-181 BID tablets — NKTR-181 tablets 100-400 mg twice daily (BID)
  Arms: NKTR-181
Drug: Placebo to match NKTR-181 BID tablets — Placebo to match NKTR-181 tablets 100-400 mg twice daily (BID)
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether a new opioid molecule, NKTR-181, is effective for the relief of moderate to severe chronic low back pain as compared to a placebo.

DETAILED DESCRIPTION:
This is an enriched enrollment, randomized withdrawal study with an open label, dose-titration period followed by a randomized, double-blind, placebo-control treatment of twelve weeks. During the double-blind treatment period, this study will evaluate the analgesic effect of NKTR-181 versus placebo in patients with moderate to severe chronic low back pain.

ELIGIBILITY:
Inclusion Criteria:

* Male or non-pregnant, non-nursing female aged 18 to 75 years old
* Clinical diagnosis of moderate to severe, chronic non-neuropathic low back pain for at least six months
* Not experiencing adequate pain relief or have failed previous treatment with non-opioid analgesics
* Opioid analgesia is necessary
* Currently taking no more than 10 mg morphine sulfate equivalents per day of short acting opioids for 14 days prior to entry
* Females of child bearing potential must be using a highly effective form of birth control. All subjects must agree to use double-barrier contraception during participation in this study and for at least 2 months after the last dose of the study drug.
* Willing and able to provide informed consent

Exclusion Criteria:

* Taking extended release or long-acting opioids within 6 months
* History of hypersensitivity, intolerance, or allergy to opioids
* Compression of spinal nerve root; spinal fracture, tumor, or abscess
* Surgical procedures on the low back in the last 12 months or facet nerve root block or radiofrequency ablation in the last 3 months
* Untreated moderate to severe sleep apnea

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1189 (Actual)
Dates: Start 2015-03-11 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2017-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (54):
- United States (54):
  - Investigator Site - Saraland, Saraland, Alabama
  - Investigator Site - Phoenix, Phoenix, Arizona
  - Investigator Site - Tempe, Tempe, Arizona
  - Investigator Site - Little Rock, Little Rock, Arkansas
  - Investigator Site - Stamford, Stamford, Connecticut
  - Investigator Site - Clearwater, Clearwater, Florida
  - Investigator Site - Fort Lauderdale, Fort Lauderdale, Florida
  - Investigator Site - Jacksonville, Jacksonville, Florida
  - Investigator Site - Orlando, Orlando, Florida
  - Investigator Site - Ormond Beach, Ormond Beach, Florida
  - Investigator Site - Plantation, Plantation, Florida
  - Investigator Site - Tampa, Tampa, Florida
  - Investigator Site - West Palm Beach, West Palm Beach, Florida
  - Investigator Site - Atlanta, Atlanta, Georgia
  - Investigator Site - Blue Ridge, Blue Ridge, Georgia
  - Investigator Site - Marietta, Marietta, Georgia
  - Investigator Site - Norcross, Norcross, Georgia
  - Investigator Site - Gurnee, Gurnee, Illinois
  - Investigator Site - West Des Moines, West Des Moines, Iowa
  - Investigator Site - Wichita, Wichita, Kansas
  - Investigator Site - Louisville, Louisville, Kentucky
  - Investigator Site - Bossier, Bossier City, Louisiana
  - Investigator Site - New Orleans, New Orleans, Louisiana
  - Investigator Site - Shreveport, Shreveport, Louisiana
  - Investigator Site - Bay City, Bay City, Michigan
  - Investigator Site - Pinconning, Pinconning, Michigan
  - Investigator Site - Biloxi, Biloxi, Mississippi
  - Investigator Site - Saint Louis 1, St Louis, Missouri
  - Investigator Site - Saint Louis 2, St Louis, Missouri
  - Investigator Site - Omaha, Omaha, Nebraska
  - Investigator Site - Las Vegas 2, Las Vegas, Nevada
  - Investigator Site - Las Vegas 1, Las Vegas, Nevada
  - Investigator Site - Rochester, Rochester, New York
  - Investigator Site - Williamsville, Williamsville, New York
  - Investigator Site - Greensboro, Greensboro, North Carolina
  - Investigator Site - Winston Salem, Winston-Salem, North Carolina
  - Investigator Site - Fargo, Fargo, North Dakota
  - Investigator Site - Beavercreek, Beavercreek, Ohio
  - Investigator Site - Cincinnati 1, Cincinnati, Ohio
  - Investigator Site - Cincinnati 2, Cincinnati, Ohio
  - Investigator Site - Columbus, Columbus, Ohio
  - Investigator Site - Duncansville, Duncansville, Pennsylvania
  - Investigator Site - Jenkintown, Jenkintown, Pennsylvania
  - Investigator Site - Rapid City, Rapid City, South Dakota
  - Investigator Site - Memphis, Memphis, Tennessee
  - Investigator Site - Arlington, Arlington, Texas
  - Investigator Site - Austin, Austin, Texas
  - Investigator Site - Killeen, Killeen, Texas
  - Investigator Site - San Antonio, San Antonio, Texas
  - Investigator Site - Salt Lake City, Salt Lake City, Utah
  - Investigator Site - West Jordan, West Jordan, Utah
  - Investigator Site - Midlothian, Midlothian, Virginia
  - Investigator Site - Norfolk, Norfolk, Virginia
  - Investigator Site - Kenosha, Kenosha, Wisconsin

REFERENCES:
- [Result] Markman J, Gudin J, Rauck R, Argoff C, Rowbotham M, Agaiby E, Gimbel J, Katz N, Doberstein SK, Tagliaferri M, Lu L, Siddhanti S, Hale M. SUMMIT-07: a randomized trial of NKTR-181, a new molecular entity, full mu-opioid receptor agonist for chronic low-back pain. Pain. 2019 Jun;160(6):1374-1382. doi: 10.1097/j.pain.0000000000001517. PMID 30747908
- See also: Related Info — https://journals.lww.com/pain/Fulltext/2019/06000/SUMMIT_07__a_randomized_trial_of_NKTR_181,_a_new.13.aspx

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First subject screened: 11Mar2015; Last subject out: 28 Dec 2016. The study was conducted at 55 medical/research sites in the United States.
Pre-assignment Details: The titration phase of the study was designed to titrate patients to a dose of NKTR-181 that provided adequate analgesia and acceptable side effects.
Groups:
- NKTR-181 (Open-label Titration Phase): NKTR-181 100-400 mg twice daily tablets
- NKTR-181 (Double-blind Treatment Phase): NKTR-181: 100-400 mg twice daily tablets
- Placebo (Double-blind Treatment Phase): Placebo: Placebo, twice daily tablets
Period: Titration Phase
Arm/Group | NKTR-181 (Open-label Titration Phase) | NKTR-181 (Double-blind Treatment Phase) | Placebo (Double-blind Treatment Phase)
Started | 1189 | 0 | 0
Completed | 610 | 0 | 0
Not Completed | 579 | 0 | 0
Period: Double-blind Maintenance Phase
Arm/Group | NKTR-181 (Open-label Titration Phase) | NKTR-181 (Double-blind Treatment Phase) | Placebo (Double-blind Treatment Phase)
Started | 0 | 309 | 301
Completed | 0 | 249 | 242
Not Completed | 0 | 60 | 59

BASELINE CHARACTERISTICS:
Groups:
- NKTR-181: NKTR-181 (Double-blind Treatment Phase)
- Placebo: Placebo (Double-blind Treatment Phase)
- Total: Total of all reporting groups
Arm/Group | NKTR-181 | Placebo | Total
Number analyzed (Participants) | 309 | 301 | 610
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.0 (12.7) | 50.7 (12.5) | 51.4 (12.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 187 | 170 | 357
  Male | 122 | 131 | 253
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3 | 3 | 6
  Asian | 4 | 2 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 2 | 2
  Black or African American | 95 | 93 | 188
  White | 205 | 196 | 401
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 2 | 4 | 6
Screening Baseline Pain Intensity in Numeric Rating Scale (NRS) [Mean (Standard Deviation); unit: units on a scale] — The pain intensity in NRS is an 11-point numerical rating scale ranging from 0 (no pain) to 10 (worst possible pain).
  Screening baseline was the 7-day average immediately prior to the first dose of NKTR-181
  units on a scale | 6.7 (0.9) | 6.8 (0.9) | 6.73 (0.9)

OUTCOME MEASURES:

1. Primary Outcome: The Change in Weekly (ie, 7-day Average) Pain Score at the End of Double-blind, Randomized Treatment Period, Relative to the Weekly Score at the End of Titration (Double-blind Baseline)
Description: The daily pain intensity is an 11-point numerical rating scale ranging from 0 (no pain) to 10 (worst possible pain).
Time Frame: 12 Weeks of randomized double blinded period
Population: The analysis set (N=610) is the intention-to-treat population, which was defined as all randomized subjects
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | NKTR-181 | Placebo
Number analyzed (Participants) | 309 | 301
units on a scale | 0.9 (0.11) | 1.5 (0.11)
Statistical Analysis 1: Comparison: NKTR-181 vs Placebo; NKTR-181 (Double-blind Treatment Phase), Placebo (Double-blind Treatment Phase); Test type: Superiority; p = 0.0019, z-test; Mean Difference (Net) = -0.55

2. Secondary Outcome: Responder Analysis Based on Percent Reduction in Pain Intensity
Description: A responder is defined by the Sponsor as a randomized subject who completes the double-blind Randomized Treatment Period and experiences improvement in the Week 12 Weekly Pain Score from Screening Pain Score. This includes the proportion of responders with at least 30% and at least 50% reduction in pain intensity.
Time Frame: Screening Baseline through Week 12
Measure: Count of Participants; unit: Participants
Arm/Group | NKTR-181 | Placebo
Number analyzed (Participants) | 309 | 301
Participants
  Subjects with 30% improvement | 220 | 172
  Subjects with 50% improvement | 158 | 114

3. Secondary Outcome: Patient Global Impression of Change (PGIC): Number of Responders
Description: The PGIC assesses the change in overall status relative to the initiation of the treatment. The scale measures global change of overall status on a 7-point scale (1 = No change (or condition has got worse), 2 = Almost the same, 3 = A little better, 4 = Somewhat better, 5 = Moderately better, 6 = Better, 7 = A great deal better). The proportion of subjects responding " A great deal better " and "better" was summarized by treatment group.
Time Frame: Screening Baseline through Week 12
Measure: Count of Participants; unit: Participants
Arm/Group | NKTR-181 | Placebo
Number analyzed (Participants) | 309 | 301
Participants | 159 | 100

4. Secondary Outcome: Change in Sleep Quality in the Medical Outcome Study Sleep Scale - Revised (MOS Sleep-R)
Description: The MOS Sleep Scale measure sleep parameters contains 12 items. Eleven of them scored using a 5-point response scale and across 5 dimensions of sleep, including disturbance (4 items), sleep problems index (9 items), somnolence (3 items), adequacy (2 items), and respiratory impairments (2 items). The original survey items are converted to a 0 to 100 range (by Converting 1 to 0, 2 to 25, 3 to 50, 4 to 75, and 5 to 100). Items in each dimension (disturbance, sleep problems index, somnolence, adequacy, respiratory impairments) of sleep are averaged together to create the score for the scale. The range of each sleep dimension is from 0 to 100. Higher score of sleep disturbance, somnolence, sleep indices, and respiratory impairments indicates relatively worse sleep problem, whereas lower scores for sleep adequacy indicate worse sleep problems.
Time Frame: Screening Baseline through Week 12
Population: The MOS Sleep-R was analyzed and presented as a change from Screening Baseline to Week 12 in double blinded treatment period. Subjects who discontinued from treatment early were not included in this analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | NKTR-181 | Placebo
Number analyzed (Participants) | 254 | 253
units on a scale
  Sleep Disturbance | -16.7 (23.9) | -9.5 (22.8)
  Sleep Problems Index | -11.6 (18.9) | -6.9 (18.4)
  Respiratory Impairments | -3.5 (18.9) | -2.2 (18.6)
  Sleep Adequacy | 9.1 (26.1) | 4.0 (25.6)
  Somnolence | -6.1 (21.0) | -7.4 (21.8)

5. Secondary Outcome: Change in Sleep Quantity Measure in Hours in the Medical Outcome Study Sleep Scale - Revised (MOS Sleep-R)
Description: The 12 items of the MOS Sleep Scale measure sleep parameters across 6 dimensions of sleep, including disturbance (4 items), sleep problems index (9 items), quantity (1 item), somnolence (3 items), adequacy (2 items), and respiratory impairments (2 items). One of the 12 items, Sleep quantity, records the actual number of hours slept. Reported here is the sleep quantity.
Time Frame: Screening Baseline through Week 12
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | NKTR-181 | Placebo
Number analyzed (Participants) | 254 | 253
hours | 0.3 (1.1) | 0.2 (1.2)

6. Secondary Outcome: Change in Roland Morris Disability Questionnaire (RMDQ)
Description: The RMDQ contains 24 items that is used to quantify the impact of low back pain on subject's ability to perform daily activities, mood and sleep. The questionnaire consists of 24 statements derived from the Sickness Impact Profile, with the addition of the phrase "because of my back." The questionnaire covers the areas of mobility, self-care, and sleeping.
  The RMDQ score is the total number of items checked which is from a minimum of 0 to a maximum of 24; the greater the score the grater the physical disability due to lower back pain.
Time Frame: Screening Baseline through Week 12
Population: The RMDQ was analyzed and presented as a change from Screening Baseline to Week 12 in double blinded treatment period. Subjects who discontinued from treatment early were not included in this analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | NKTR-181 | Placebo
Number analyzed (Participants) | 254 | 253
units on a scale | -4.0 (5.7) | -3.5 (5.6)

ADVERSE EVENTS:
Time Frame: Adverse events were reported starting immediately after the subject provided written informed consent through the end of study, which is approximately 20 to 25 weeks for each subject.
Description: Adverse events were collected after the subject provided written informed consent till the end of study through spontaneous reports or were observed during other assessments. All ongoing AEs were followed until resolution or for 14 days after the subject's last visit, whichever came first. All SAEs were followed until resolution, stabilization of condition, return to baseline, or until follow-up is no longer possible.
Groups:
- NKTR-181 (Titration Phase); NKTR-181 (Double-blind Treatment Phase): NKTR-181 100-400 mg twice daily tablets
- Placebo (Double-blind Treatment Phase): Placebo, twice daily tablets
Arm/Group | NKTR-181 (Titration Phase) | NKTR-181 (Double-blind Treatment Phase) | Placebo (Double-blind Treatment Phase)
Serious Adverse Events (participants affected / at risk) | 9/1189 | 5/309 | 6/301
Other Adverse Events (participants affected / at risk) | 803/1189 | 111/309 | 66/301
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | NKTR-181 (Titration Phase) (N=1189) | NKTR-181 (Double-blind Treatment Phase) (N=309) | Placebo (Double-blind Treatment Phase) (N=301)
Atrial Fibrillation (Cardiac disorders) | 1 | 0 | 0
Blindness transient (Eye disorders) | 1 | 0 | 0
Large intestine perforation (Gastrointestinal disorders) | 1 | 0 | 0
Diverticulum intestinal (Gastrointestinal disorders) | 0 | 0 | 1
Chest Pain (General disorders) | 0 | 1 | 0
Cellulitis (Infections and infestations) | 1 | 0 | 0
Gastrointestinal infection (Infections and infestations) | 1 | 0 | 0
Herpes virus infection (Infections and infestations) | 1 | 0 | 0
Infective exacerbation of chronic obstructive airways (Infections and infestations) | 1 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 0
Diverticulitis (Infections and infestations) | 0 | 1 | 0
Bacterial infection (Infections and infestations) | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 0 | 1
Rib fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Skin abrasions (Injury, poisoning and procedural complications) | 0 | 0 | 1
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 1 | 0 | 0
Dysarthria (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Renal failure (Renal and urinary disorders) | 0 | 1 | 0
Angiodema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Hypertension (Vascular disorders) | 0 | 1 | 0
Malignant hypertension (Vascular disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | NKTR-181 (Titration Phase) (N=1189) | NKTR-181 (Double-blind Treatment Phase) (N=309) | Placebo (Double-blind Treatment Phase) (N=301)
Constipation (Gastrointestinal disorders) | 425 | 27 | 9
Nausea (Gastrointestinal disorders) | 176 | 32 | 18
Vomiting (Gastrointestinal disorders) | 67 | 15 | 5
Dry mouth (Gastrointestinal disorders) | 66 | 7 | 1
Diarrhoea (Gastrointestinal disorders) | 35 | 8 | 17
Fatigue (General disorders) | 61 | 4 | 1
Somnolence (Nervous system disorders) | 107 | 8 | 1
Headache (Nervous system disorders) | 83 | 10 | 14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If a joint manuscript has not been submitted for publication within twelve (12) months of completion or termination of the study, the PI is free to publish separately, upon provision of any proposed publication or manuscript to the Sponsor at least sixty (60) days before it is submitted or otherwise disclosed.